CLINICAL TRIAL: NCT01127854
Title: Pilot Study to Evaluate the Contribution of Gene Variants to Idiopathic Urolithiasis
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivan E. Porter, II, Principal Investigator, Mayo Clinic
Other Study IDs: 09-007826
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones; Urolithiasis; Calcium Oxalate Urolithiasis
Keywords: kidney stone; urolithiasis; calcium oxalate kidney stone; calcium oxalate stone; calcium oxalate
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis, Calcium Oxalate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Urine and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases
- Controls

SUMMARY:
Recent investigations from this group have identified that genetic variants of genes associated with monogenic forms of nephrolithiasis are expressed in idiopathic calcium oxalate kidney stone patients and could influence stone forming risk. Utilizing patient samples from the Mayo Clinic Florida Kidney Stone Registry, we will demonstrate that expression of these heterozygous mutations in idiopathic nephrolithiasis act as genetic modifiers of disease presentation increasing risk of kidney stone formation. Complimented by the analysis of environmental and lifestyle risk factors, these studies will define environmental and genetic susceptibility factors involved in kidney stone formation and reoccurrence.

DETAILED DESCRIPTION:
Nephrolithiasis occurs in approximately 1 in 10 individuals in the United States with increasing prevalence noted over the past three decades (ref: Worcester E, Coe F. Nephrolithiasis. Prim Care Clin Office Pract 35 (2008) 369-391). Recurrence is common - occurring in more than 50% of these patients, many of whom require surgical intervention. An estimated 5-6 billion dollars a year is spent on the treatment of kidney stones. Symptoms of kidney stones include flank pain, blood in the urine, and nausea and vomiting. Beyond acute attacks associated with considerable morbidity and cost, recent reports have identified an association between kidney stone formation and an increased risk for the development of hypertension, chronic kidney disease, end stage renal disease and myocardial infarction. Therefore, nephrolithiasis not only impacts socioeconomics but also has broader public health implications. Genetic and environmental risk factors have both been linked to nephrolithiasis with about 40% of the patients presenting with kidney stones having at least one relative who is also a stone former. Genetic variants that are causative of monogenic forms of nephrolithiasis have been well defined. However the frequency of these monogenic mutations and their presence as predisposing factors of disease is poorly understood within the idiopathic stone forming population.

We recently identified that heterozygous mutations of HOGA1, a gene that is associated with the onset of primary hyperoxularia Type III, are also present within the idiopathic stone forming population and absent in matched controls. These findings suggest that the presence of these mutations could be indicative of an increased risk for kidney stone formation within these patients. We therefore propose to; Aim 1: Validate and expand our previous studies to define that genetic variations of HOGA1 are a predisposing factor for idiopathic calcium-oxalate stone formation, and Aim 2: Mutational analysis of genes involved in kidney stone formation for determination of genetics of risk. These clinical studies will identify the frequency of known genetic variants associated with monogenic forms of nephrolithiasis within idiopathic stone forming populations and associate their presence with heightened risk. Patient genomic DNA, blood, clinical data and risk data are available from the Mayo Clinic Florida Kidney Stone Registry. Genomic DNA and RNA will be assessed for mutations within HOGA1 and their significance as predisposing factors for disease evaluated through statistical analysis and compared to environmental factors for risk. Evaluations will also be undertaken in control patient samples, identifying that these mutations are specific for idiopathic kidney stone formation risk. Furthermore, genetic variants within AGXT, GRHPR, HOGA1, CLCN5, OCRL1, SLC3A1, SLC7A9, and APRT will be analyzed for frequency in idiopathic nephrolithiasis patients and control patient populations to determine their role as predictive genetic markers for idiopathic disease risk.

This proposed study has the potential to identify genetic variants that are predisposing factors for idiopathic kidney stone formation and are predictive of disease risk. These studies have relevance to personalized treatment regimens for disease intervention and targeted prevention of reoccurrence. Furthermore, the knowledge gained pertaining to genetic variants in idiopathic stone formers may lead to the creation of genetic tests for the early diagnosis of those patients at higher risk of idiopathic nephrolithiasis.

Nine hundred idiopathic kidney stone formers and 900 non-kidney stone forming controls will be examined for the evaluation of HOGA1 genetic variants. We propose to use the patient resources provided by the Kidney Stone Registry and control samples from the Mayo Clinic BioBank in Florida. Briefly, for the Kidney Stone Registry, all cases presenting with kidney stones are invited to enroll in the Registry. Enrolled patients are approached for data abstraction, risk factor questionnaire completion, biospecimen collection (blood and DNA) and long-term follow-up. At this time we have over 1500 phenotypically well characterized patients enrolled within the registry with approximately 500 new patient enrollments each year. For these studies, we will only utilize samples and patient histories from idiopathic calcium oxalate stone formers and controls. The PI of this application oversees the running of this registry. Controls will be selected from patients who have consented genomic DNA samples to the Mayo Clinic Biobank (http://mayoresearch.mayo.edu/mayo/research/biobank/). These controls are defined as patients who have a negative personal history of symptomatic urolithiasis and no family history of kidney stone formation. Dr. Parker oversees the running of the Mayo Clinic BioBank in Florida. Patient records and information will only be available to the PI, co-investigator and biostatistician named on this proposal. Phenotypical Analysis: Phenotype data will be extracted from patient's medical records. All patients provide informed consent to DNA testing and record review under research protocols approved by the Mayo Clinic Institutional Review Board. Risk Factor Data Collection: A self-administered questionnaire is provided to each patient on their initial visit by the practitioner, is provided within the Appendix. Those patients that have consented to be enrolled in the Kidney Stone Registry and consented to be included in this study will be our case study group. The questionnaire requests patients to provide information pertaining to family history, lifestyle and environmental risk factors for kidney stone formation. All questionnaires are reviewed by the study coordinator for completeness and accuracy of responses.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* History of calcium oxalate stones
* 18 years of age or older
* Willing to provide a blood sample, and questionnaire

Controls:

* 18 years of age or older
* No personal history of urolithiasis
* Willing to provide a blood sample and questionnaire

Exclusion Criteria:

Cases:

* Secondary causes of urolithiasis including: Bowel disease, Renal tubular acidosis, hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic in Jacksonville, FL
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2009-12; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To identify the frequency of known genetic variants associated with monogenic forms of nephrolithiasis within idiopathic stone forming populations and associate their presence with heightened risk. | December 2018

CONTACTS AND LOCATIONS:
Overall Officials: William E Haley, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials